CLINICAL TRIAL: NCT04173806
Title: Development and Evaluation of an Online Telemedicine Course Through Facebook: a Randomized Controlled Trial
Brief Title: Evaluation of an Online Telemedicine Course Through Facebook
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Cender Udai Quispe Juli, Principal Investigator, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 104043
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2019-11

CONDITIONS: Telemedicine; Training
Keywords: Education, Medical; Online Social Networking; Computer User Training; Telemedicine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facebook group (Experimental): Participants will be included in an online classroom through a "closed group" of Facebook to receive an asynchronous course of telemedicine.
  Interventions: Other: Facebook intervention
- Control group (Active Comparator): In this group the participants are exposed to the same course of telemedicine but on the Moodle educational platform.
  Interventions: Other: Control Training:

INTERVENTIONS:
Other: Facebook intervention — The intervention consists of the content of the course on telemedicine through a "closed group" of Facebook according to the established syllabus whose educational material is video classes, discussion forums and online questionnaires. The duration of the course will be 5 weeks, each week two classes will be uploaded to the Facebook platform in succession until the course is completed. So that the student can visualize the content progressively and continuously.
  Arms: Facebook group
Other: Control Training: — In this group the participants are exposed to the same course content and perform similar activities as the intervention group on Facebook during the same period but on the Moodle educational platform. The Moodle platform was chosen because it has been widely used in several institutions, with a large user community worldwide, with approximately 50,000 registrations in more than 200 countries and due to the many easy-to-use educational tools it offers. So it is one of the educational platforms that has demonstrated its efficiency in the medical educational field.
  Arms: Control group

SUMMARY:
Health professionals with adequate training are required to provide quality remote care. There are few telemedicine and telehealth training programs for doctors and medical students. On the other hand, the use of social networks (Facebook and Twitter) as a medical education tool is becoming frequent. However, there is a lack of conclusive evidence in terms of its effectiveness. The objective of the present study is to develop and evaluate a telemedicine course for resident doctors through Facebook and compare it with one through Moodle. A randomized, triple-blind, parallel block controlled trial will be conducted that tests the effectiveness of an educational intervention through Facebook compared to another control intervention using Moodle. Intervention training is a telemedicine course focused on teleconsultation provided through Facebook. Control training is the same educational content but through Moodle. The level of telemedicine knowledge of the participants before and after the intervention will be evaluated. The inferential analysis to see the association between the variables of interest will be carried out by Student's T tests or analysis of variance (ANOVA). If potential confounding factors were found, the variable will be adjusted through linear regression. The pre and post intervention analysis will be carried out with student t or wilcoxon rank test according to the normality of the data. Resident doctors who receive the telemedicine course through Facebook are expected to have a greater knowledge gain than those who take the course through Moodle.

DETAILED DESCRIPTION:
Main Objective:

Develop and evaluate a telemedicine course for resident doctors through Facebook and compare it with one through Moodle.

Study Design:

A randomized, triple-blind, parallel block controlled trial will be conducted that tests the effectiveness of an educational intervention through Facebook compared to another control intervention using Moodle. Intervention training is a telemedicine course focused on teleconsultation provided through Facebook. Control training is the same educational content but through Moodle. The level of telemedicine knowledge of the participants before and after the intervention will be evaluated. In addition, at the end of the intervention the level of satisfaction of the participants will be evaluated.

Population:

Resident doctors of the Faculty of Medicine of the Universidad Peruana Cayetano Heredia.

Sample:

In a previous study, the response within each group of subjects was normally distributed with a standard deviation of 2.62. If the true difference in the experimental and control means is 3, the investigators will have to study 13 experimental subjects and 13 control subjects to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with the probability (power) 0.8. The probability of Type I error associated with this test of this null hypothesis is 0.05. Then the investigators consider the 30% follow-up loss rate, according to previous reports, our final sample size being 38 people, therefore our intervention and control group will be made up of 19 people each. This is the minimum sample size needed; however, a larger number improves the power of the study.

Group assignment:

Participants will be randomly assigned to the intervention or control training by simple random assignment (random numbers generated by computer). Once the assigned group of each participant has been determined, they will be given access to the course content on their respective platforms.

Ethical considerations:

This project will be guided by the principles of scientific integrity. The project was submitted to the Institutional Committee of Research Ethics of the Universidad Peruana Cayetano Heredia for evaluation and approval. The content of the classes (educational videos) will be based on specialized scientific literature and current technical standards. In the end of the course, participants will have received telemedicine training as part of their curriculum and they will increase their professional skills. They will not be offered any additional incentive. When enrolling in the course, participants will be informed of the research objectives and procedures. Resident doctors will accept the use of their data generated by the course for the purpose of this study voluntarily

ELIGIBILITY:
Inclusion Criteria:

* Physician enrolled in the resident program of Universidad Peruana Cayetano Heredia, who has passed the first year of residence.
* Motivation to learn telemedicine and participate in educational activities during the intervention.
* Access to the internet through a computer or mobile device during the intervention of the study.

Exclusion Criteria:

* Resident doctors who have had some type of training in e-Health, telemedicine or telehealth.
* Rotating doctors from other national or foreign universities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-08-29 (Estimated)

PRIMARY OUTCOMES:
Level of Knowledge about telemedicine | through study completion, an average of 1 month
  Measured by automatic scoring after the participant took the tests on a web platform. The instrument is a questionnaire made up of 32 multiple-choice questions about knowledge in telemedicine focused on teleconsultation. The test is according to guidelines of the National Board of Medical Examiners of the United States. Each correct question is worth 3.125 points so the scale range will be 0-100 points in total but then it will be converted to vigesimal score from 0 to 20 points, being the passing grade 11.00.

SECONDARY OUTCOMES:
The satisfaction assessment will be carried out through the Wang questionnaire (Likert scale) | through study completion, an average of 1 month
  Wang questionnaire is an electronic learning satisfaction model of 26 elements related to four qualities: content, learning interface, personalization, learning community and also with two questions which refer to the overall measurement in the context of end-user satisfaction. The measurement scale will be a 7-point Likert scale, with scores ranging from 1 to 7 ("strongly disagree" to "strongly agree" respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Cender U Quispe Juli, MD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Universidad Peruana Cayetano Heredia, Medicine School, Lima, San Martín de Porres, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuckson RV, Edmunds M, Hodgkins ML. Telehealth. N Engl J Med. 2017 Oct 19;377(16):1585-1592. doi: 10.1056/NEJMsr1503323. No abstract available. PMID 29045204
- [Background] Celes RS, Rossi TRA, de Barros SG, Santos CML, Cardoso C. [Telehealth as state response strategy: systematic reviewLa telesalud como estrategia de respuesta del Estado: revision sistematica]. Rev Panam Salud Publica. 2018 Aug 10;42:e84. doi: 10.26633/RPSP.2018.84. eCollection 2018. Portuguese. PMID 31093112
- [Background] Pathipati AS, Azad TD, Jethwani K. Telemedical Education: Training Digital Natives in Telemedicine. J Med Internet Res. 2016 Jul 12;18(7):e193. doi: 10.2196/jmir.5534. PMID 27405323
- [Background] van Galen LS, Wang CJ, Nanayakkara PWB, Paranjape K, Kramer MHH, Car J. Telehealth requires expansion of physicians' communication competencies training. Med Teach. 2019 Jun;41(6):714-715. doi: 10.1080/0142159X.2018.1481284. Epub 2018 Jun 26. PMID 29944031
- [Background] Edirippulige S, Armfield NR. Education and training to support the use of clinical telehealth: A review of the literature. J Telemed Telecare. 2017 Feb;23(2):273-282. doi: 10.1177/1357633X16632968. Epub 2016 Jul 8. PMID 26892005
- [Background] dos Santos Ade F, Alves HJ, Nogueira JT, Torres RM, Melo Mdo C. Telehealth distance education course in Latin America: analysis of an experience involving 15 countries. Telemed J E Health. 2014 Aug;20(8):736-41. doi: 10.1089/tmj.2013.0291. Epub 2014 Jun 5. PMID 24901742
- [Background] Nicolai L, Schmidbauer M, Gradel M, Ferch S, Anton S, Hoppe B, Pander T, von der Borch P, Pinilla S, Fischer M, Dimitriadis K. Facebook Groups as a Powerful and Dynamic Tool in Medical Education: Mixed-Method Study. J Med Internet Res. 2017 Dec 22;19(12):e408. doi: 10.2196/jmir.7990. PMID 29273572
- [Background] Ghanem O, Logghe HJ, Tran BV, Huynh D, Jacob B. Closed Facebook groups and CME credit: a new format for continuing medical education. Surg Endosc. 2019 Feb;33(2):587-591. doi: 10.1007/s00464-018-6376-9. Epub 2018 Aug 13. PMID 30105596
- [Background] Pander T, Pinilla S, Dimitriadis K, Fischer MR. The use of Facebook in medical education--a literature review. GMS Z Med Ausbild. 2014 Aug 15;31(3):Doc33. doi: 10.3205/zma000925. eCollection 2014. PMID 25228935
- [Background] Ellaway R, Masters K. AMEE Guide 32: e-Learning in medical education Part 1: Learning, teaching and assessment. Med Teach. 2008 Jun;30(5):455-73. doi: 10.1080/01421590802108331. PMID 18576185
- [Background] Masters K, Ellaway R. e-Learning in medical education Guide 32 Part 2: Technology, management and design. Med Teach. 2008 Jun;30(5):474-89. doi: 10.1080/01421590802108349. PMID 18576186